CLINICAL TRIAL: NCT03819855
Title: External Validation of the RESAS (REnnes Septic Arthritis Score) Septic Arthritis Prognosis Score in an Acute Arthritis Cohort of Less Than 30 Days
Brief Title: External Validation of a Septic Arthritis Prognosis Score
Acronym: SYNOLACTATES +
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_30015_SYNOLACTATES-PLUS
Record Dates: First submitted 2019-01-11; First posted 2019-01-29 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study

DETAILED DESCRIPTION:
Septic arthritis is a diagnostic emergency for acute arthritis because it is accompanied by an excess of mortality of 11% and frequent functional sequelae in about 50% of cases in the year. However, it remains rare with an estimated annual incidence of 1 to 5/100000, and a prevalence of about 10% in front of an acute arthritis table sent to an emergency department.

The diagnosis is based on the bacteriological culture which finds the presence of a microorganism within the joint. However, only 80% of septic arthritis is bacteriologically documented due to low inoculum, the presence of fragile bacteria (Neisseria sp) or especially untimely antibiotherapy prior to joint puncture.

In addition, the bacteriological culture takes an average of 3 days to become positive, which may delay the implementation of appropriate antibiotic therapy.

It is therefore essential that the clinician can rely on other clinical or biological parameters, reliable and fast for better diagnostic orientation.

A first study: SYNOLACTATES showed the interest of the measurement of glucose and synovial lactate for the diagnosis of septic arthritis with very good performances. A RESAS score (REnnes Septic Arthritis Score) was constructed from these results to assess the likelihood of septic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Any acute arthritis less than or equal to 30 days;
* Achievement of a joint puncture in routine care as part of the diagnostic assessment of this acute arthritis;
* Affiliation to a social security scheme;
* No one opposes his participation in the research.

Exclusion Criteria:

* Age below 18 years;
* Major persons subject to legal protection (safeguard of justice, guardianship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients performing joint puncture in routine care as part of a diagnostic assessment of acute arthritis
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
RESAS (Rennes Septic Arthritis Score) | Up to 3 days (time to collect laboratory results)
  Composite score of 4 biological variables of the synovial liquid (macroscopically purulent liquid and/or Synovial White Cells Counts (SWCC) ≥ 75000/mm3, synovial crystal vizualization, synovial lactate dosage, synovial glucose dosage). Each variable is weighted as follows: macroscopically purulent liquid or SWCC ≥ 75000/mm3 (+3 points), UMS (-4 points) or CPP (-2 points) crystal Vizualization, lactate ≥ 11.5 mmol/L (+6 points) or 10-11.4 mmol/L (+4 points) or 8.5-9.9 mmol/L (+2 points), glucose ≤ 1.0 mmol/L (+4 points), 1.1-1.8 mmol/L (+2 points), yielding a total between -4 and 13.

SECONDARY OUTCOMES:
Macroscopic synovial fluid appearance | Up to 1 day (time to collect clinical parameters)
  Expressed in multiple qualitative variable: purulent, trouble, clear citrine appearance, hemarthrosis or clear with blood threads
Microscopic synovial analysis | Up to 3 days (time to collect laboratory results)
  Presence of crystals in synovial fluid: urate monosodic (UMS) crystal (Yes or No), and calcium pyrophosphate crystal (CPP) (Yes or No)
Synovial White Cells Count (SWCC) | Up to 3 days (time to collect laboratory results)
  Number (n) of White cells in synovial fluid. (quantitative variable expressed in n/mm3)
Total lactates, D-lactate, glucose | Up to 3 days (time to collect laboratory results)
  Measures of total lactate, D-lactate et glucose in synovial fluid (quantitative variable expressed in mmol/L)
Others synovial proteic markers | Up to 3 days (time to collect laboratory results)
  Measures of CRP (mg/L) in synovial fluid
Others synovial proteic markers | Up to 3 days (time to collect laboratory results)
  Measures of Procalcitonine (ng/mL) in synovial fluid
Others synovial proteic markers | Up to 3 days (time to collect laboratory results)
  Measures of Calprotectin (ng/mL) in synovial fluid
Multielemental analysis by ICP-MS | Up to 3 days (time to collect laboratory results)
  Screening multielemental in synovial fluid
Number of classical clinical marker (quantitative variable) to diagnosis of septic arthritis | Up to 1 day (time to collect clinical parameters)
  Fever (expressed in Celcius degree)
Number of classical clinical marker (quantitative variable) to diagnosis of septic arthritis | Up to 1 day (time to collect clinical parameters)
  Duration of symptoms (expressed in day)
Number of classical clinical marker (qualitative variable) to diagnosis of septic arthritis | Up to 1 day (time to collect clinical parameters)
  Co-morbidity promoting infection (diabetes, cirrhosis, HIV, severe chronic renal failure, rheumatoid arthritis, other inflammatory rheumatic diseases, immunosuppressive treatments such as corticosteroids, conventional synthetic-DMARDs, biological-DMARDs) (Yes or No)
Number of classical clinical marker (qualitative variable) to diagnosis of septic arthritis | Up to 1 day (time to collect clinical parameters)
  Number of joints affected (Ordinal variable)
Parameters that may influence the bacteriological results of synovial fluid | Up to 1 day (time to collect clinical parameters)
  NSAIDs, corticosteroids, antibiotics within 15 days of joint puncture (qualitative variable: Yes or No)
Number of hospitalization potentially avoided by the early elimination of an arthritis diagnosis and their cost, from the point of view of illness insurance | Date of hospitalization until 2 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Coiffier, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France